CLINICAL TRIAL: NCT04863807
Title: A Retrospective Review of Rib Fracture Pain Management at a London Major Trauma Centre Comparing Erector Spinae Plane Blocks, Serratus Anterior Plane Blocks and Epidurals
Brief Title: A Retrospective Review of Rib Fracture Pain Management at a London Major Trauma Centre
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19SM5668; 276933 (Other: HRA and Health and Care Research Wales (HCRW))
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Rib Fractures; Pain, Acute
Keywords: epidural; erector spinae block; serratus anterior block
MeSH Terms: conditions — Rib Fractures; Acute Pain | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Thoracic epidural for rib fracture management: Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years that meet the criteria for the Imperial College Healthcare National Health Service (NHS) Trust 'Invasive rib fracture management pathway'
  Interventions: Procedure: Regional Anaesthesia
- Erector Spinae block for rib fracture management: Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years that meet the criteria for the Imperial College Healthcare NHS Trust 'Invasive rib fracture management pathway'
  Interventions: Procedure: Regional Anaesthesia
- Serratus Anterior block for rib fracture management: Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years that meet the criteria for the Imperial College Healthcare NHS Trust 'Invasive rib fracture management pathway'
  Interventions: Procedure: Regional Anaesthesia

INTERVENTIONS:
Procedure: Regional Anaesthesia — Thoracic epidural/Erector Spinae block/Serratus Anterior block

SUMMARY:
Thoracic epidural analgesia (TEA) is widely considered to be the current gold standard treatment for rib fracture pain and is used in the Imperial invasive treatment pathway for rib fractures. However, TEA are often contraindicated due to other injuries or the use of anticoagulant medications, which also contraindicates other invasive nerve block techniques e.g. paravertebral catheters. A number of case reports have reported the safe use of alternative techniques such as Serratus Anterior Blocks (SAPB) and Erector Spinae Blocks (ESPB) and the anaesthesia community has taken them up widely based on this relatively limited evidence. In view of this, Womack et al recently published a large retrospective review examining the safety and efficacy of ultrasound guided paravertebral catheter analgesia techniques in rib fracture management along with small numbers of ESPBs. However, this data did not report the analgesic efficacy, patient reported pain relief or respiratory complications.The goal is to advance this body of evidence by reviewing our larger data set concerning the use of TEA and alternative regional techniques such as ESPB and SAPB. This comprehensive review will benefit patients by documenting the efficacy and safety of these techniques for clinicians managing rib fracture patients.

DETAILED DESCRIPTION:
Primary Objective The primary objective is to examine whether novel fascial plane blocks, e.g. SAPB and ESPB, are effective pain relief modalities in patients with rib fractures - the proportion of patients with a reduction in pain.

Secondary Objectives

The investigators review the safety profile and complications of TEA and alternative analgesic techniques such as ESPB and SAPB used for rib fracture management in our trauma centre. In particular the effects of regional anaesthesia techniques on:

1. Opioid use
2. Nausea & vomiting
3. Respiratory complications
4. Intubation & non-invasive ventilation (NIV)
5. ICU admission for respiratory complications

The investigators will assess the duration of use and complication profile of regional anaesthetic techniques, including infection, analgesic failure and damage to other structures during insertion e.g. the lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years
* Meet the criteria for the Imperial College Healthcare NHS Trust 'Invasive rib fracture management pathway'

Exclusion Criteria:

* Under 18 years old
* Prisoners
* Pregnant
* Private patients
* Meet the criteria for the Imperial College Healthcare NHS Trust 'Non-invasive rib fracture management pathway'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years
  * Meet the criteria for the Imperial College Healthcare NHS Trust 'Invasive rib fracture management pathway' (see Appendix A)
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boyne Bellew, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperiial Collge Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon BJ, Cushman J, Barraco R, Lane V, Luchette FA, Miglietta M, Roccaforte DJ, Spector R; EAST Practice Management Guidelines Work Group. Pain management guidelines for blunt thoracic trauma. J Trauma. 2005 Nov;59(5):1256-67. doi: 10.1097/01.ta.0000178063.77946.f5. No abstract available. PMID 16385313
- [Background] Jones KM, Reed RL 2nd, Luchette FA. The ribs or not the ribs: which influences mortality? Am J Surg. 2011 Nov;202(5):598-604. doi: 10.1016/j.amjsurg.2010.09.029. Epub 2011 Aug 26. PMID 21872207
- [Background] Adhikary SD, Liu WM, Fuller E, Cruz-Eng H, Chin KJ. The effect of erector spinae plane block on respiratory and analgesic outcomes in multiple rib fractures: a retrospective cohort study. Anaesthesia. 2019 May;74(5):585-593. doi: 10.1111/anae.14579. Epub 2019 Feb 10. PMID 30740657
- [Result] Ahn Y, Gorlinger K, Alam HB, Eikermann M. Pain-associated respiratory failure in chest trauma. Anesthesiology. 2013 Mar;118(3):701-8. doi: 10.1097/ALN.0b013e318283996b. No abstract available. PMID 23403516
- [Result] Barnea Y, Kashtan H, Skornick Y, Werbin N. Isolated rib fractures in elderly patients: mortality and morbidity. Can J Surg. 2002 Feb;45(1):43-6. PMID 11837920
- [Result] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Result] Womack J, Pearson JD, Walker IA, Stephens NM, Goodman BA. Safety, complications and clinical outcome after ultrasound-guided paravertebral catheter insertion for rib fracture analgesia: a single-centre retrospective observational study. Anaesthesia. 2019 May;74(5):594-601. doi: 10.1111/anae.14580. Epub 2019 Jan 27. PMID 30687939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Records will be identified by searching the Trauma Audit and Research Network database, routinely collected database of all patients admitted with traumatic injury within the Imperial College Healthcare Trust. The study will be conducted from 11/11/2020 until the 31/01/2023. We plan to review rib injured patient's electronic notes that have received these interventions from January 2016 until December 2019 and categorise the information for analysis as set out in study outcomes.
Period: Overall Study
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Started | 325 | 26 | 38
Completed | 325 | 26 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management | Total
Number analyzed (Participants) | 325 | 26 | 38 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 166 | 7 | 12 | 185
  >=65 years | 159 | 19 | 26 | 204
Age, Continuous [Median (Full Range); unit: years] | 63 [19 to 97] | 76 [37 to 98] | 69 [26 to 95] | 66 [19 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 8 | 18 | 133
  Male | 218 | 18 | 20 | 256
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 325 | 26 | 38 | 389

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With a Reduction in Pain
Description: The investigators will review pain scores as recorded by clinical staff over 72 hours to assess pain relief efficacy, A verbal rating scale classifying pain as mild, moderate or severe is used at Imperial Data from the acute pain round records will also provide details regarding breathing comfort levels of the patient, coughing ability and deep inspiratory effort. These are recorded as yes/no answers and the team will assess the proportion of patients showing a reduction in pain scores.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
Participants | 101 | 6 | 15

2. Secondary Outcome: Opioid Consumption (mg/24h)
Description: Data regarding type of opiate use
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: 24hr opioid consumption (mg)
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
24hr opioid consumption (mg) | 0 [0 to 7.9] | 15 [3.1 to 41.8] | 10 [0 to 18.8]

3. Secondary Outcome: Nausea and Vomiting
Description: The incidence of nausea in the 72 hours post block will be recorded with the number of episodes in each patient
Time Frame: 72 hours post block
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
Participants | 117 | 10 | 2

4. Secondary Outcome: Number of Patients With Respiratory Complication(s)'
Description: Lower respiratory tract infections: defined as raised CRP/ White Cell Count, new consolidation on CXR or antibiotics being started at clinician discretion.
  Empyema or parapneumonic effusions: defined as radiological evidence of fluid collections within the pleural space and therapeutic interventions required for treatment e.g. aspiration and drainage.
Time Frame: Length of stay up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
Participants | 110 | 10 | 13

5. Secondary Outcome: Intensive Care Admission
Description: ICU admission for respiratory complications, number of days of mechanical ventilation.
Time Frame: Length of stay up to 8 weeks in days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
Participants | 44 | 2 | 6

6. Secondary Outcome: Intensive Care Admission
Description: Number of patients requiring intubation and ventilation
Time Frame: Length of stay up to 8 weeks in days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
Participants | 30 | 1 | 2

7. Secondary Outcome: Number of Days of Mechanical Ventilation
Description: Number of days of mechanical ventilation for patients undergoing Intensive care mechanical ventilation
Time Frame: Length of stay up to 8 weeks in days
Measure: Median (Full Range); unit: days
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
Number analyzed (Participants) | 325 | 26 | 38
days | 0 [0 to 45] | 0 [0 to 11] | 0 [0 to 9]

ADVERSE EVENTS:
Time Frame: Duration of hospital admission
Description: 389 participants were included, 6 patients had >1 block during their inpatient stay but did not affect their participation in the trial and/or the collection of results, therefore 389 patients.
Arm/Group | Thoracic Epidural for Rib Fracture Management | Erector Spinae Block for Rib Fracture Management | Serratus Anterior Block for Rib Fracture Management
All-Cause Mortality (participants affected / at risk) | 9/325 | 2/38 | 3/26
Serious Adverse Events (participants affected / at risk) | 206/325 | 14/26 | 22/38
Other Adverse Events (participants affected / at risk) | 0/325 | 0/26 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thoracic Epidural for Rib Fracture Management (N=325) | Erector Spinae Block for Rib Fracture Management (N=26) | Serratus Anterior Block for Rib Fracture Management (N=38)
ICU admission for respiratory complication (Respiratory, thoracic and mediastinal disorders) | 66 | 3 | 7
Intubation & Mechanical Ventilation (Respiratory, thoracic and mediastinal disorders) | 30 | 1 | 2
Any lung complication (Respiratory, thoracic and mediastinal disorders) | 110 | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04863807/Prot_SAP_000.pdf